CLINICAL TRIAL: NCT06408610
Title: Moderate Continuous Versus High Interval Intensity Training on Gut Dysbiosis and Glucagon Like Peptide Hormone in Irritable Bowel Syndrome
Brief Title: Moderate Continuous Versus High Interval Intensity Training on Gut Dysbiosis and GLP1 Hormone in IBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Marwa Saeed Salama, PhD candidate, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: P.T./REC/012/004224
Record Dates: First submitted 2024-05-07; First posted 2024-05-10 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Irritable Bowel Syndrome; Obesity; Dysbiosis
MeSH Terms: conditions — Irritable Bowel Syndrome; Obesity; Dysbiosis | interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: 1. Patients will receive moderate intensity continuous training (MICT)
  2. Patients will receive high intensity interval training (HIIT)
  3. Patients will be instructed to follow low fermentable short chain carbohydrates diet (low FODMAP)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- moderate intensity continuous training (Experimental): Patients will receive moderate intensity continuous training The program will be in form of Frequency Moderate continues training will be scheduled 3 times per week for 12 weeks Intensity 65-75% of target heart rate.
  Duration 40 minutes per session.
  Interventions: Other: moderate intensity continuous training
- high intensity interval training (Experimental): Patients will receive high intensity interval training. The program will be in form of Frequency: High intensity interval training will be scheduled 3 times per week for 12 week Intensity 90% of target heart rate including 10 bouts of 1 minute interspersed with 10 bouts of 1 minute of active recovery 50% of target heart rate. Duration the session will last 30 minutes includes warming up and cooling down periods.
  Interventions: Other: moderate intensity continuous training
- low fermentable short chain carbohydrates diet (Experimental): Patients will be instructed to follow low fermentable short chain carbohydrates diet (low FODMAP) intervention for 12 weeks limiting daily fermented carbohydrate and dairy products and increase intake of protein, whole grains, fruits and vegetables
  Interventions: Other: moderate intensity continuous training

INTERVENTIONS:
Other: moderate intensity continuous training — exercise and diet
  Other Names: high intensity interval training; low fermentable short chain carbohydrates diet (low FODMAP)

SUMMARY:
investigating the response of gut bacteria via measuring short chain fatty acids and Glucagon like peptide hormone to two different modes of exercises in pre-diabetic, obese patients with irritable bowel syndrome. It will be hypothesized that there will be no significant difference between the moderate continuous versus high interval intensity training on gut dysbiosis and glucagon like peptide hormone in irritable bowel syndrome.

DETAILED DESCRIPTION:
The human gastrointestinal tract represents one of the largest organ between the host, environmental factors and antigens in the human body. In an average life time, around 60 tonnes of food pass through the human GI tract, along with an abundance of microorganisms from the environment which impose a huge threat on gut integrity. The collection of bacteria, archaea and eukarya colonising the GI tract is termed the 'gut microbiota' and has co-evolved with the host over thousands of years to form an intricate and mutually beneficial relationship.The gut microbiota enjoys a mutualistic relationship with the host, harvesting additional energy and nutrients from the diet and protecting the host from pathogens. The resident bacteria produce a wide range of metabolites and chemicals that influence host function and these include short-chain fatty acids such as butyrate, which is essential for the integrity of the colonic epithelium.

However, there is potential for these mechanisms to be disrupted as a result of an altered microbial composition, known as dysbiosis. Human Gut dysbiosis is linked to many pathologic conditions disturbing the energy metabolism; such as obesity and atherosclerosis. The microbiota in the human gut is mostly composed of bacterial phyla: Firmicutes and Bacteroidetes. Firmicutes bacteria are Gram-positive one. It plays a key role in the nutrition and metabolism of the host through SCFA synthesis. Through their metabolic products, Firmicutes bacteria are indirectly connected with other tissues and organs and regulate hunger and satiety. In contrast, Bacteroidetes bacteria are Gram negative and associated with immunomodulation. Increased or decreased Firmicutes / Bacteroidetes (F/B) ratio are associated with the development of obesity or irritable bowel disease (IBD). Short-chain fatty acids (SCFAs), the primary metabolite for colonocytes, are produced in the intestinal lumen by commensal anaerobic bacteria via carbohydrate fermentation. they play a role in preserving gut barrier functions, and have immunomodulatory and anti-inflammatory properties also it regulates the synthesis of the hunger-suppressing hormones leptin, peptide YY, and glucagon- like peptide 1. The gut microbiota can also affect appetite and satiety via vagus nerve activation or immune-neuroendocrine mechanisms. Irritable bowel syndrome (IBS) is a common gastrointestinal disorder characterized by chronic abdominal pain and changes in bowel habits without any known organic causes. Fecal SCFAs abnormalities have been reported in patients with IBS, implying that alterations in SCFAs might be related to IBS. The cause of IBS remains unknown, and no single treatment is found to be universally applicable to all patients with IBS. Among humans, positive correlations were reported between bacterial diversity, butyrate-producing bacteria and cardiorespiratory fitness (VO2max), and higher turnover of carbohydrates and proteins, and concentrations of short-chain fatty acids in athletes compared to sedentary controls. There is also growing evidence that physical activity status and exercise training may shape the gut microbiome.

Physical activity stimulates bacterial community richness by altering SCFAs-producing species, as well as favoring the colonization of health and athletic performance-promoting strains. The ability to promote a bacterial composition capable of protecting the intestinal mucosa also it was found that the effects on gut microbiome seem to gradually disappear when the physical activity is no longer practiced. Moderate aerobic exercise affects the intestinal system mainly through gut immune function gut barrier integrity through tight junction proteins expression and IgA production hypothalamic-pituitary-adrenal (HPA) axis stimulation which, in turn, affects enteric nervous system and intestinal transit time, as well as gut motility, intestinal pH and gut hormones release and bile acids metabolism within enterohepatic circulation. High intensity interval training (HIIT) encompasses exercise prescriptions that are tailored to individual needs and can be used in most any exercise setting. This ability to adapt makes HIIT a valuable tool in the exercise programming of patients with a chronic disease. HIIT has a positive effect on the Bacteroidetes/Firmicutes ratio and also increased the alpha diversity in gut microbiota.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index must be 30-34.9 kg\m
* Clinical diagnosis of irritable bowel syndrome
* Must be Pre-diabetic HbA1c of 5.7 - 6.4.
* Must be sedentary subject

Exclusion Criteria:

* Communication disorders
* Gasterointestinal bleeding
* Antibiotics or probiotics in the last 2 months
* Recent surgeries in the last 6 months
* Colorectal cancer or any terminal diseases
* Fibromylgia or Multiple sclerosis
* Palpable abdominal mass
* Cardiovascular diseases
* Active smokers
* Musculoskeletal injuries that interfere with exercise program
* Upper respiratory infections
* Uncontrolled hypertension

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-05-17 (Actual)

PRIMARY OUTCOMES:
Short Chain fatty acids | before the start of the trial and at the end of the trial 3 months
  fecal sample will be separated. Applying four analytes, including total SCFAs, acetate, propionate, and butyrate, will be targeted. Final concentrations will be calculated based on internal standards and are expressed as micromoles per gram of wet feces (μmol/g). Techniques and predictive approaches will be used across. gas chromatography will be used to quantify Short Chain Fatty Acids (SCFAs) from fecal samples
Glucagon like peptide hormone | before the start of the trial and at the end of the trial 3 months
  Glucagon like peptide hormone will be measure with Elisa Kit an Enzyme-Linked Immunosorbent Assay. The plate will be pre-coated with Human GLP-1 antibody

SECONDARY OUTCOMES:
Body Mass Index | before the start of the trial and at the end of the trial 3 months
  weight and height will be recorded to calculate body mass index (BMI) according to the following equation BMI= weight/height2 (Kg/m2)
irritable bowel syndrome severity scoring system | before the start of the trial and at the end of the trial 3 months
  This five-item questionnaire will measure IBS symptom severity by addressing abdominal pain (frequency and severity), bloating, dissatisfaction with bowel habits, and interference with daily activities. Each question score ranges from 0 to 100 and a higher score indicates more severe GI symptoms. A total score of 75-175 represents mild IBS, 176-300 moderate IBS and >300 severe IBS
rritable bowel syndrome quality of life questionnaire | before the start of the trial and at the end of the trial 3 months
  The IBS-QoL is a condition-specific instrument will be used to assess the impact of IBS and effects of treatment. It consists of 34 questions which cover eight domains including dysphoria, interference with activity, body image, health worry, food avoidance, social reaction, sexual, and relationships. Each item has a five-point response scale (not at all, slightly, moderately, quite a bit, extremely).
  The responses are summed and averaged for a total score and transformed to a scale between 0 and 100: higher scores indicating better IBS-specific QoL

CONTACTS AND LOCATIONS:
Overall Officials: Donia M Elmasry, Doctorate, Study Director — Faculty of physiotherapy Cairo University
Locations (2):
- Egypt (2):
  - Faculty of medicine cairo university, Cairo
  - Faculty of physiotherapy cairo university, Giza

IPD SHARING:
Plan to Share IPD: Yes
study protocol and final results
Supporting Information: Study Protocol, ICF
Time Frame: May 2024 till March 2025
Access Criteria: Researchers

REFERENCES:
- [Background] Aziz I, Simren M. The overlap between irritable bowel syndrome and organic gastrointestinal diseases. Lancet Gastroenterol Hepatol. 2021 Feb;6(2):139-148. doi: 10.1016/S2468-1253(20)30212-0. Epub 2020 Nov 13. PMID 33189181
- [Background] Cataldi S, Poli L, Sahin FN, Patti A, Santacroce L, Bianco A, Greco G, Ghinassi B, Di Baldassarre A, Fischetti F. The Effects of Physical Activity on the Gut Microbiota and the Gut-Brain Axis in Preclinical and Human Models: A Narrative Review. Nutrients. 2022 Aug 11;14(16):3293. doi: 10.3390/nu14163293. PMID 36014798
- [Background] Cella V, Bimonte VM, Sabato C, Paoli A, Baldari C, Campanella M, Lenzi A, Ferretti E, Migliaccio S. Nutrition and Physical Activity-Induced Changes in Gut Microbiota: Possible Implications for Human Health and Athletic Performance. Foods. 2021 Dec 10;10(12):3075. doi: 10.3390/foods10123075. PMID 34945630
- [Background] Chen L, Sun X, Khalsa AS, Bailey MT, Kelleher K, Spees C, Zhu J. Accurate and reliable quantitation of short chain fatty acids from human feces by ultra high-performance liquid chromatography-high resolution mass spectrometry (UPLC-HRMS). J Pharm Biomed Anal. 2021 Jun 5;200:114066. doi: 10.1016/j.jpba.2021.114066. Epub 2021 Apr 6. PMID 33866297
- [Background] Clark T, Morey R, Jones MD, Marcos L, Ristov M, Ram A, Hakansson S, Franklin A, McCarthy C, De Carli L, Ward R, Keech A. High-intensity interval training for reducing blood pressure: a randomized trial vs. moderate-intensity continuous training in males with overweight or obesity. Hypertens Res. 2020 May;43(5):396-403. doi: 10.1038/s41440-019-0392-6. Epub 2020 Jan 14. PMID 31937915
- [Background] DeGruttola AK, Low D, Mizoguchi A, Mizoguchi E. Current Understanding of Dysbiosis in Disease in Human and Animal Models. Inflamm Bowel Dis. 2016 May;22(5):1137-50. doi: 10.1097/MIB.0000000000000750. PMID 27070911
- [Background] Denou E, Marcinko K, Surette MG, Steinberg GR, Schertzer JD. High-intensity exercise training increases the diversity and metabolic capacity of the mouse distal gut microbiota during diet-induced obesity. Am J Physiol Endocrinol Metab. 2016 Jun 1;310(11):E982-93. doi: 10.1152/ajpendo.00537.2015. Epub 2016 Apr 26. PMID 27117007
- [Background] Elhosseiny D, Mahmoud NE, Manzour AF. Factors associated with irritable bowel syndrome among medical students at Ain Shams University. J Egypt Public Health Assoc. 2019 Dec 4;94(1):23. doi: 10.1186/s42506-019-0023-8. PMID 32813140
- [Background] Gupta AK, Maity C. Efficacy and safety of Bacillus coagulans LBSC in irritable bowel syndrome: A prospective, interventional, randomized, double-blind, placebo-controlled clinical study [CONSORT Compliant]. Medicine (Baltimore). 2021 Jan 22;100(3):e23641. doi: 10.1097/MD.0000000000023641. PMID 33545934
- [Background] Koh A, De Vadder F, Kovatcheva-Datchary P, Backhed F. From Dietary Fiber to Host Physiology: Short-Chain Fatty Acids as Key Bacterial Metabolites. Cell. 2016 Jun 2;165(6):1332-1345. doi: 10.1016/j.cell.2016.05.041. PMID 27259147
- [Background] Kuhre RE, Wewer Albrechtsen NJ, Hartmann B, Deacon CF, Holst JJ. Measurement of the incretin hormones: glucagon-like peptide-1 and glucose-dependent insulinotropic peptide. J Diabetes Complications. 2015 Apr;29(3):445-50. doi: 10.1016/j.jdiacomp.2014.12.006. Epub 2014 Dec 15. PMID 25623632
- [Background] Lin L, Zhang J. Role of intestinal microbiota and metabolites on gut homeostasis and human diseases. BMC Immunol. 2017 Jan 6;18(1):2. doi: 10.1186/s12865-016-0187-3. PMID 28061847
- [Background] Mohammed AA, Moustafa HA, Nour-Eldein H, Saudi RA. Association of anxiety-depressive disorders with irritable bowel syndrome among patients attending a rural family practice center: a comparative cross-sectional study. Gen Psychiatr. 2021 Dec 13;34(6):e100553. doi: 10.1136/gpsych-2021-100553. eCollection 2021. PMID 34970639
- [Background] Monda V, Villano I, Messina A, Valenzano A, Esposito T, Moscatelli F, Viggiano A, Cibelli G, Chieffi S, Monda M, Messina G. Exercise Modifies the Gut Microbiota with Positive Health Effects. Oxid Med Cell Longev. 2017;2017:3831972. doi: 10.1155/2017/3831972. Epub 2017 Mar 5. PMID 28357027
- [Background] Portincasa P, Bonfrate L, Vacca M, De Angelis M, Farella I, Lanza E, Khalil M, Wang DQ, Sperandio M, Di Ciaula A. Gut Microbiota and Short Chain Fatty Acids: Implications in Glucose Homeostasis. Int J Mol Sci. 2022 Jan 20;23(3):1105. doi: 10.3390/ijms23031105. PMID 35163038
- [Background] Prince SA, Cardilli L, Reed JL, Saunders TJ, Kite C, Douillette K, Fournier K, Buckley JP. A comparison of self-reported and device measured sedentary behaviour in adults: a systematic review and meta-analysis. Int J Behav Nutr Phys Act. 2020 Mar 4;17(1):31. doi: 10.1186/s12966-020-00938-3. PMID 32131845
- [Background] Resende AS, Leite GSF, Lancha Junior AH. Changes in the Gut Bacteria Composition of Healthy Men with the Same Nutritional Profile Undergoing 10-Week Aerobic Exercise Training: A Randomized Controlled Trial. Nutrients. 2021 Aug 18;13(8):2839. doi: 10.3390/nu13082839. PMID 34444999
- [Background] Rettedal EA, Cree JME, Adams SE, MacRae C, Skidmore PML, Cameron-Smith D, Gant N, Blenkiron C, Merry TL. Short-term high-intensity interval training exercise does not affect gut bacterial community diversity or composition of lean and overweight men. Exp Physiol. 2020 Aug;105(8):1268-1279. doi: 10.1113/EP088744. Epub 2020 Jun 17. PMID 32478429
- [Background] Shukohifar M, Mozafari Z, Rahmanian M, Mirzaei M. Performance of body mass index and body fat percentage in predicting metabolic syndrome risk factors in diabetic patients of Yazd, Iran. BMC Endocr Disord. 2022 Aug 31;22(1):216. doi: 10.1186/s12902-022-01125-0. PMID 36045359
- [Background] Singh R, Zogg H, Wei L, Bartlett A, Ghoshal UC, Rajender S, Ro S. Gut Microbial Dysbiosis in the Pathogenesis of Gastrointestinal Dysmotility and Metabolic Disorders. J Neurogastroenterol Motil. 2021 Jan 30;27(1):19-34. doi: 10.5056/jnm20149. PMID 33166939
- [Background] Song BK, Kim YS, Kim HS, Oh JW, Lee O, Kim JS. Combined exercise improves gastrointestinal motility in psychiatric in patients. World J Clin Cases. 2018 Aug 16;6(8):207-213. doi: 10.12998/wjcc.v6.i8.207. PMID 30148149
- [Background] Stojanov S, Berlec A, Strukelj B. The Influence of Probiotics on the Firmicutes/Bacteroidetes Ratio in the Treatment of Obesity and Inflammatory Bowel disease. Microorganisms. 2020 Nov 1;8(11):1715. doi: 10.3390/microorganisms8111715. PMID 33139627
- [Background] Sun Q, Jia Q, Song L, Duan L. Alterations in fecal short-chain fatty acids in patients with irritable bowel syndrome: A systematic review and meta-analysis. Medicine (Baltimore). 2019 Feb;98(7):e14513. doi: 10.1097/MD.0000000000014513. PMID 30762787
- [Background] Thursby E, Juge N. Introduction to the human gut microbiota. Biochem J. 2017 May 16;474(11):1823-1836. doi: 10.1042/BCJ20160510. PMID 28512250
- [Background] Varney J, Barrett J, Scarlata K, Catsos P, Gibson PR, Muir JG. FODMAPs: food composition, defining cutoff values and international application. J Gastroenterol Hepatol. 2017 Mar;32 Suppl 1:53-61. doi: 10.1111/jgh.13698. PMID 28244665
- [Background] Wang L, Alammar N, Singh R, Nanavati J, Song Y, Chaudhary R, Mullin GE. Gut Microbial Dysbiosis in the Irritable Bowel Syndrome: A Systematic Review and Meta-Analysis of Case-Control Studies. J Acad Nutr Diet. 2020 Apr;120(4):565-586. doi: 10.1016/j.jand.2019.05.015. Epub 2019 Aug 28. PMID 31473156

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-11-30): https://cdn.clinicaltrials.gov/large-docs/10/NCT06408610/Prot_SAP_ICF_001.pdf